CLINICAL TRIAL: NCT04230616
Title: Comparison of Clinical Outcome and Alignment of NAVIO Total Knee Arthroplasty and Conventional Total Knee Arthroplasty A Prospective, Randomized, Controlled, Single Blind Study
Brief Title: Efficacy and Safety of NAVIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sint-Trudo Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S63149
Record Dates: First submitted 2020-01-08; First posted 2020-01-18 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2020-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional total knee arthroplasty (Active Comparator): conventional total knee arthroplasty with standard intramedullary alignment guide
  Interventions: Procedure: total knee arthroplasty; Radiation: CT scan
- NAVIO total knee arthroplasty (Active Comparator): NAVIO assisted total knee arthroplasty
  Interventions: Procedure: total knee arthroplasty; Radiation: CT scan

INTERVENTIONS:
Procedure: total knee arthroplasty — total knee arthroplasty
Radiation: CT scan — The first 52 participants will recieve a pre- and postoperative CT scan of the hip, knee and ankle.

SUMMARY:
The goal of the study is to compare the efficacy, safety and costs of the NAVIO™ system with the conventional intramedullary alignment guide for total knee replacement in a clinical setting. The hypothesis is that total knee arthroplasty (TKA) with the use of NAVIO™ is at least as efficient and safe as TKA with the use of conventional intramedullary alignment guiding.

ELIGIBILITY:
Inclusion Criteria:

* Painful and disabled knee joint resulting from osteoarthritis where one or more compartments are involved, as assessed by X-ray
* High need to obtain pain relief and improve function
* Above 18 years old
* Able and willing to follow instructions
* Informed consent

Exclusion Criteria:

* Active infection in knee
* General infection
* Failure of previous joint replacement
* Post-operative or post traumatic malalignment of the knee/leg
* Pregnancy
* Not able or willing to undergo CT-scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Difference in planned and achieved alignment in degrees based on CT scan pre- and postoperatively (first 52 participants) | within 6 weeks pre-surgery and 6 weeks post-surgery
  Difference in preoperatively planned and postoperatively achieved alignment of both the femoral and tibial component of the prosthesis in the frontal, sagittal and coronal plane. Deviations (in degrees varus/valgus, flexion extension, and internal/external rotation) from calculated positions (of both components) to bony anatomic landmarks, used by NAVIO to align the prosthesis, will be obtained.
Difference in planned and achieved mechanical axis in degrees based on CT scan pre- and postoperatively (first 52 participants) | within 6 weeks pre-surgery and 6 weeks post-surgery
  Preoperatively planned and postoperatively achieved mechanical axis of the operated leg. The mechanical axis is defined as the angle between a line from the centre of rotation of the hip to the centre of the femoral component and a line from the centre of the tibial plateau to the centre of the ankle.
Difference in percentage of outliers of alignment on CT scan pre- and postoperatively (first 52 participants) | within 6 weeks pre-surgery and 6 weeks post-surgery
  Percentage of outliers in alignment (defined as > 3 degrees deviation from positions calculated by software) of the femoral and tibial components in frontal, sagittal and transverse plane.
Difference in percentage of outliers of mechanical axis based on CT scan pre- and postoperatively (first 52 participants) | within 6 weeks pre-surgery and 6 weeks post-surgery
  Percentage of outliers (defined as > 3 degrees deviation from neutral) in mechanical axis of the of the operated leg. The mechanical axis is defined as the angle between a line from the centre of rotation of the hip to the centre of the femoral component and a line from the centre of the tibial plateau to the centre of the ankle.
Mean change in the visual analogue scale scores | within 6 weeks preoperative, 24 hours post-surgery, day of discharge, 6 weeks post-surgery, 3 months post-surgery, 1 year post-surgery, 2 years post-surgery, 5 years post-surgery, 10 years post-surgery
  Comparison is made between the two study arms, a higher visual analogue pain score means a worse outcome
Mean change in the American Knee Society Score | within 6 weeks preoperative, 3 months post-surgery, 1 year post-surgery, 2 years post-surgery, 5 years post-surgery, 10 years post-surgery
  in a total of 50 points, stability, 25 points, and range of motion, 25 points. The maximum score of 100 points . Comparison is made between the two study arms. A higher American Knee Society Score means a better outcome
Mean change in the Oxford Knee Score | within 6 weeks preoperative, 3 months post-surgery, 1 year post-surgery, 2 years post-surgery, 5 years post-surgery, 10 years post-surgery
  Comparison is made between the two study arms, score between 0 and 48. Better score means better outcome
Mean change in the Lower Extremities Activity scale | within 6 weeks preoperative, day of discharge, 6 weeks post-surgery, 3 months post-surgery, 1 year post-surgery, 2 years post-surgery, 5 years post-surgery, 10 years post-surgery
  Comparison is made between the two study arms, score between 0 and 80. The minimal clinically important difference is 9 scale points. The lower the score the greater the disability.
Mean change in the The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | within 6 weeks preoperative, 3 months post-surgery, 1 year post-surgery, 2 years post-surgery, 5 years post-surgery, 10 years post-surgery
  Comparison is made between the two study arms. Five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). The higher the score, the poorer the function
Difference in mechanical axis of the prosthesis between the two study arms based on Long-leg X-rays | within 6 weeks preoperative, 6 weeks post-surgery, 1 year post-surgery, 5 years post-surgery, 10 years post-surgery
  Post-operative (at 6 week visit) the baseline mechanical axis will be measured as the angle between a line connecting the center of the femoral head with the center of the knee and the line connecting the center of the knee with the center of the ankle.
Difference in positioning of the prosthesis between the two study arms based on Long-leg X-rays | within 6 weeks preoperative, 6 weeks post-surgery, 1 year post-surgery, 5 years post-surgery, 10 years post-surgery
  In order to measure positioning of the prosthesis (coronal alignment), long-leg, weight-bearing, standing anteroposterior and lateral X-rays will be made
Difference in wear between the two study arms based on Long-leg X-rays | within 6 weeks preoperative, 6 weeks post-surgery, 1 year post-surgery, 5 years post-surgery, 10 years post-surgery
  In the long term, wear can be roughly measured by measuring again the mechanical axis of the leg and comparing this with baseline mechanical axis and by measuring the distance between medial and lateral femoral condyles and medial and lateral tibial platform respectively.
Significant difference in length of hospital stay between the two study arms | 1 day of discharge from the hospital
  Length of hospital stay (in days) will be registered for both groups.
Operation Time | intraoperative (Time will be recorded from the moment of incision until bandage is being placed)
  Compare the duration of surgery between the two study arms
Significant difference in blood loss between study arms | Intra-operatively until 24 hours post-surgery. .
  Blood loss will be measured intra-operatively and up to 24 hours post-operatively.
  The amount of rinsing liquid will be subtracted from the total amount collected in the suction device to obtain the amount (ml) of intra-operative blood loss. The weight of grids and compresses will be measured post-operatively and dry weight will be subtracted from this value to obtain blood loss not collected in the suction device (1mg = 1ml).
  On day 2 post-operative, Hb and Ht will obtained.
Difference in adverse events | through study completion, an average of 10 years
  Complication registration will be done throughout the entire study period
Difference in frequency of infection | through study completion, an average of 10 years
  When infection is present, this will be noted on the complication registry form and appropriate action will be taken. Distinction will be made between superficial infections and deep infections.
Difference in frequency of trombo-embolic complications | through study completion, an average of 10 years
  Attention will be focused on clinical signs of deep vein thrombosis and pulmonary embolism.
Difference in frequency of wound problems | From day of surgery until 5 days post-surgery
  Persistent wound leakage will be registered. Persistent leakage is defined as leakage lasting 5 days after surgery.
Difference in frequency of loosening | through study completion, an average of 10 years.
  Loosening of tibial or femoral components of the prosthesis as seen on X-ray.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bollars, Dr., Principal Investigator — Orthopedic Association Sint-Trudo Hospital
Locations (1):
- Orthopaedic Association Sint-Trudo Hospital, Sint-Truiden, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: Undecided